CLINICAL TRIAL: NCT04423848
Title: Supportive Oncology Care at Home Intervention for Patients With Lymphoma
Brief Title: Home Hospital for Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume due to poor accrual.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-613
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma
Keywords: Lymphoma; Home Care Services, Hospital-Based; Cancer Care
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Hospital for Lymphoma (Experimental): The Home Hospital for Lymphoma intervention entails the following: patient-reported symptoms and vital signs with appropriate triggers for phone calls and home visits, and regular communication with oncology clinicians regarding care delivered at home to ensure continuity of care.
  Interventions: Other: Home Hospital for Lymphoma

INTERVENTIONS:
Other: Home Hospital for Lymphoma — Remote monitoring and home-based care designed for hospitalized patients with lymphoma

SUMMARY:
The goal of this research is to evaluate an intervention, which the investigators call "Home Hospital for Lymphoma," that involves remote patient monitoring and home-based supportive care for patients hospitalized with lymphoma at Massachusetts General Hospital.

DETAILED DESCRIPTION:
This research study is a single arm pilot Feasibility Study, which is the first-time investigators are examining this hospital at home intervention for patients with lymphoma.

The research study procedures include screening for eligibility, questionnaires, remote patient monitoring (e.g. patient-reported symptoms and home monitored vital signs) and home-based supportive care (e.g. visits to patients' homes to address and manage any concerning issues identified), and interviews of participants, caregivers, and clinicians asking their perceptions of the Home Hospital for Lymphoma program.

Participants will include 3 groups:

Enrolled participants receiving the hospital at home intervention, caregivers of participants, and clinicians.

Participants will be in the research study for about six months after consent. It is expected that up to 38 participants will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Receiving their lymphoma care with curative intent at MGH (treatment intent based upon chemotherapy order in the electronic medical record)
* Hemodynamically stable during the first 24 hours of hospital admission at MGH
* Residing within the designated geographic area for MGH Home Hospital Service (an approximately 10-mile radius from MGH)
* Able to communicate and respond to questionnaires in English
* Lives with a family member or a friend who supports the patient at home
* Deemed eligible for supportive oncology care at home based on the MGH Home Hospital clinician evaluation

Exclusion Criteria:

* Those admitted to the intensive care unit
* Have high oxygen requirement (FIO2 > 0.4)
* Experience active angina or cardiac arrythmias
* Have a planned inpatient surgical or interventional procedure
* Have uncontrolled psychiatric illness or impaired cognition that prohibits complying with the study procedures
* Have uncontrolled pain requiring intravenous pain medications
* Those deemed ineligible based on the Home Hospital Service clinician evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
enrollment rate | 1 year
  The primary endpoint is feasibility. The proposed intervention will be deemed feasible if at least 60% of eligible patients are enrolled in the study
retention rate | 1 year
  The primary endpoint is feasibility. The proposed intervention will be deemed feasible if those enrolled patients complete at least 60% of daily patient-reported symptom assessment.

SECONDARY OUTCOMES:
Acceptability of the intervention | 1 year
  Qualitative acceptability ratings from patients, caregivers, and clinicians obtained via exit individual interviews regarding acceptability (i.e. usefulness, effectiveness, and relevance of the intervention) from patients, family caregivers, and clinicians. The intervention will be deemed acceptable if ≥ 60% of patients, family caregivers, and clinicians report that the intervention was helpful.
Rates of completion of daily vital signs | 1 year
  Proportion of participants that complete daily reporting of vital signs during their home hospital admission.
Rates of Adverse Events | 1 year
  The rates of Adverse Events and Serious Adverse Events that are judged by the treating lymphoma clinician to be at least possibly related to the study intervention.

OTHER OUTCOMES:
Symptom burden (Edmonton Symptom Assessment System-revised - ESAS-r) | 1 year
  Change in participants' symptom burden as measured by the ESAS-r throughout the study. The ESAS-r ranges 0-10 for each symptom with higher scores indicating worse symptom burden.
Psychological distress (Hospital Anxiety and Depression Scale - HADS) | 1 year
  Change in psychological distress as measured by the HADS, with subscale ranges from 0-21 with higher scores indicating worse psychological distress.
Quality of life (Functional Assessment of Cancer Therapy-General - FACT-G) | 1 year
  Change in quality of life as measured by the FACT-G throughout the study, with range of 0-108 and higher scores indicating better quality of life.
Length of home hospital admission | 1 year
  Number of days the participant receives home hospital care through the home hospital program.
Number of home visits | 1 year
  Number of home visits required, their average duration, the issues addressed at home, and the interventions delivered to participants at their home.
Number of phone calls | 1 year
  Number of phone calls required per participants as well as the average duration of these calls.
Number of urgent visits | 1 year
  The number of urgent visits to clinic per participant and the proportion of participants who have an urgent visit to clinic.
Number of emergency department (ED) visits The number of imaging tests ordered during home hospital admission | 1 year
  The number of emergency department (ED) visits per participant and the proportion of participants who have an ED visit.
Number of hospital readmissions | 1 year
  The number of hospital readmissions in 30 days per participant and the proportion of participants who have a hospital readmission within 30 days.
Number of imaging studies | 1 year
  The number of imaging studies obtained per participant during the Home Hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation